CLINICAL TRIAL: NCT04267653
Title: Lactoferrin Efficacy Versus Ferrous Sulfate in Treatment of Patients With Iron Deficiency Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gaber Ahmed, pediatrician, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17100915
Record Dates: First submitted 2020-02-05; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Iron Deficiency Anemia Treatment
Keywords: Iron deficiency anemia; Lactoferrin; Ferrous sulfate
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lactoferrin (Active Comparator): Oral bovine lactoferrin (bfl) 100 mg once daily on empty stomach
  Interventions: Drug: Lactoferrin Bovine
- ferrous sulfate (Active Comparator): Oral ferrous sulfate 3-6 mg/kg of elemental iron/day in divided doses
  Interventions: Drug: Ferrous Sulfate
- combined (Active Comparator): combined therapy (both lactoferrin and ferrous sulfate)
  Interventions: Drug: Lactoferrin Bovine; Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: Lactoferrin Bovine — treatment for 30 days
  Other Names: Pravotin sachet
  Arms: combined; lactoferrin
Drug: Ferrous Sulfate — treatment for 30 days
  Other Names: ferrovit syrup
  Arms: combined; ferrous sulfate

SUMMARY:
Lactoferrin (Lf) is a mammalian cationic iron binding glycoprotein belonging to the transferrin family which was discovered 70 years ago, and isolated simultaneously from human and bovine milks in 1960. It is widely distributed in all biological fluids and is also expressed by immune cells, which release it under stimulation by pathogens

ELIGIBILITY:
Inclusion Criteria:all patients with iron deficiency anemia from 2 to 15 years old

-

Exclusion Criteria:

* Anemia rather than iron deficiency anemia.
* Family history of blood disease.
* Patients with thalassemia trait.
* Patients with chronic illness.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
comparison of efficacy of lactoferrin versus ferrous sulfate tharapy in treatment of patients with iron deficiency anemia. | 30 days
  Complete blood count will be done before and after therapy to detect the effect of the therapy on serum hemoglobin(g/d)
Comparison of efficacy of lactoferrin versus ferrous sulfate tharapy in treatment of patients with iron deficiency anemia. | 30 days
  Total serum iron(ug/d) will be done before and after therapy to detect effect of the therapy on total serum iron level (ug/d)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gaber Ahmed, Principal Investigator — Assiut University
Locations (1):
- AssuitU, Asyut, Egypt